CLINICAL TRIAL: NCT01242735
Title: Testing the Efficacy of an Exercise Intervention for Patients With OCD
Brief Title: Exercise and Health Intervention for Patients With Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1006-001; 1R01MH086513-01A1 (NIH)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; OCD; Exercise; Aerobic Exercise
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Motor Activity | interventions — Exercise; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): 12-week moderate-intensity behavioral exercise intervention (AE)
  Interventions: Behavioral: Aerobic exercise
- Health and Wellness (Active Comparator): 12-week health and wellness education control (HEC)
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Aerobic exercise — 12-week moderate-intensity behavioral exercise intervention. Weekly sessions with an exercise physiologist who will also assign weekly exercise goals.
  Arms: Exercise
Behavioral: Health and Wellness — 12-week health and wellness education control. Weekly sessions about 12 different topics related to OCD, led by an OCD expert.
  Arms: Health and Wellness

SUMMARY:
The purpose of this study is to test the effect of a moderate-intensity aerobic exercise intervention for Obsessive Compulsive Disorder (OCD) patients interested in reducing symptoms. The investigators expect that this project will contribute much needed knowledge about the role that aerobic exercise can play in managing the effects of OCD. If moderate-intensity aerobic exercise is efficacious in helping individuals with OCD manage obsessions and compulsions, this will establish that aerobic exercise may be a valuable adjunct to other OCD treatments such as medication and therapy.

ELIGIBILITY:
Inclusion Criteria:

1. are between 18 and 65 years of age
2. are sedentary, i.e. have not participated in regular aerobic physical exercise for at least 90 minutes per week during the past three months
3. currently engaged in at least 12 weeks of stable dose pharmacotherapy and/or are currently engaged in cognitive-behavioral therapy for the past 13 weeks
4. meet Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria for OCD as assessed by the Structured Clinical Interview for DSM Disorders, Patient Version (SCID-P)
5. have Y-BOCS score greater than 16

Exclusion Criteria:

1. DSM-IV diagnosis of substance abuse/dependence except for nicotine dependence
2. DSM-IV diagnosis of anorexia or bulimia nervosa
3. DSM-IV diagnosis of bipolar disorder
4. history of psychotic disorder or current psychotic symptoms
5. current suicidality or homicidality
6. marked organic impairment
7. physical or medical problems that would not allow for safe exercise participation
8. current pregnancy or intent to become pregnant during the next 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS; OCD symptomatology) | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Abrantes, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Szuhany KL, Steinberg MH, McLaughlin NCR, Mancebo MC, Brown RA, Greenberg BD, Simon NM, Abrantes AM. Predictors of Long-Term Exercise Engagement in Patients With Obsessive-Compulsive Disorder: The Role of Physical Activity Enjoyment. Behav Ther. 2023 Jul;54(4):610-622. doi: 10.1016/j.beth.2022.12.010. Epub 2023 Jan 5. PMID 37330252